CLINICAL TRIAL: NCT02772263
Title: Pilot Project: Community Health Assessment Program Through Emergency Medical Services
Acronym: CHAP-EMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14 210
Record Dates: First submitted 2016-05-03; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus
Keywords: Paramedicine; Community Paramedic; Elderly
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHAP-EMS Intervention (Experimental): Participants guided through a 15-20 minute defined risk assessment by a trained paramedic. Risk factors assessed were those related to cardiovascular and diabetes risk (blood pressure, diabetes-risk status, lifestyle factors), and potential for falls. Based on these, the paramedic provided education and developed an individualized action plan directing participants to use available community resources to assist them in addressing their risk factors. They were advised to return to CHAP-EMS sessions regularly for BP monitoring and follow-up. Each participant's information was faxed to his/her family physician once a month.
  Interventions: Other: CHAP-EMS

INTERVENTIONS:
Other: CHAP-EMS — The CHAP-EMS program is a low cost community program that is designed to assess community dwelling seniors for lifestyle risk factors that may impact their health and well-being and to provide targeted education to address the pertinent risk factors. Each participant is guided through a structured health-risk assessment focused on diabetes, cardiovascular disease and other potential health issues. The assessment is conducted by a trained paramedic in a common area within the community housing building. Data gathered are used to develop individualized action plans concerning health-risk reduction, to direct participants to local health activities or resources, educate on promoting health and to transmit this information to a participants' family physician.

SUMMARY:
Older adults living in subsidized housing report poorer health. Their low income and age make it harder for them to use community services. Many older adults have heart disease and diabetes, which lead to frequent emergency calls and hospital admissions. To decrease the costs of treating heart disease and diabetes through emergency and hospitalization, improved screening and health education is needed. The Community Health Assessment Program through Emergency Medical Services (CHAP-EMS) program will take place in communal areas within housing buildings of older adults and deliver a heart disease, diabetes, and falls risk check-up with health education. This is expected to improve the health of older adults leading to fewer emergency calls and hospital visits.

Paramedics on modified duties (e.g. injured) will conduct weekly, one-on-one drop-in sessions for seniors in a common area of one subsidized apartment building in Hamilton, Ontario.

DETAILED DESCRIPTION:
The CHAP-EMS research team has created a multifaceted intervention (cardiovascular, diabetes, and falls risk assessment with health education/promotion and appropriate referral) in partnership with Hamilton Paramedic Service, City Housing Hamilton (CHH), and the Community Care Access Center (CCAC) that focuses on issues experienced by older adults that often lead to EMS calls. CHAP-EMS is based on the Cardiovascular Health Awareness Program (CHAP) model, which combined individual- and population-level strategies for primary prevention and 'closed the loop' by linking participants to follow-up care. Literature demonstrates that the CHAP program resulted in a significant 9% relative reduction in admissions due to stroke, heart failure, and heart attacks in people aged 65 and over.

The original CHAP program was run by trained volunteers. This modified program will be run by accommodated paramedics (unable to assume traditional paramedic duties due to personal limitations such as pregnancy or injuries). Subsidized housing buildings house frail, seriously ill and potentially unstable individuals who may require immediate assistance. Paramedics are an excellent fit to deal with these emergent situations since their training prepares them to accurately assess the patient's health status and the environmental context, and connect patients with primary care physicians, visiting nurses, and community services including falls prevention; these skills can be expanded to provide non-urgent health care services and health promotion work. EMS administrators indicate that there is no shortage of accommodated staff at the Hamilton Paramedic Service and work considered as light duties is scarce.

The objectives are to evaluate whether a weekly 8-hour CHAP-EMS program is associated with changes in (1) number of emergency (911) EMS calls from the seniors' residence building, (2) mean blood pressure (BP) of participants and (3) diabetes risk profile of participants after one year of implementation.

ELIGIBILITY:
Inclusion Criteria:

* Living in intervention building
* Aged 65 or over

Exclusion Criteria:

* Not living in intervention building
* Under aged 65

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in rate of EMS calls over 1 year | Baseline and 1 year
  Building-level change in EMS call rate (pre-post intervention)

SECONDARY OUTCOMES:
Change in systolic and diastolic blood pressure over 1 year | Baseline and after each assessment (up to 1 year)
  Since the participants are invited to attend the intervention weekly, but are not required to attend, the number of assessments and time of assessments will vary. Multilevel analysis will be conducted that accounts for this variance in repeated measures.
Change in Canadian Diabetes Risk (CANRISK) score over 1 year | Baseline and 1 year
  The CANRISK tool provides a 10-year risk of diabetes score and will be administered by the paramedic during the CHAP-EMS session.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarwal, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal G, Angeles R, Pirrie M, Marzanek F, McLeod B, Parascandalo J, Dolovich L. Effectiveness of a community paramedic-led health assessment and education initiative in a seniors' residence building: the Community Health Assessment Program through Emergency Medical Services (CHAP-EMS). BMC Emerg Med. 2017 Mar 9;17(1):8. doi: 10.1186/s12873-017-0119-4. PMID 28274221